CLINICAL TRIAL: NCT04433481
Title: Efficacy and Safety of Dabigatran in Patients With Cirrhosis and Portal Vein Thrombosis-A Randomized Placebo Controlled Trial
Brief Title: Efficacy and Safety of Dabigatran in Patients With Cirrhosis and Portal Vein Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-30
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Liver Cirrhosis; Portal Vein Thrombosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Dabigatran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DABIGATRAN (Experimental): 150mg BD for 12 months
  Interventions: Drug: Dabigatran
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dabigatran — T. Dabigatran 150 mg twice a day
  Arms: DABIGATRAN
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
A randomized controlled trial to study the efficacy and safety of Dabigatran in Cirrhotic patients who develop PVT.In this study the patients who meet the inclusion criteria will be randomized to either receive Dabigatran or placebo [multivitamin tablet]. Blood samples will be taken &Imaging will be done accordingly to notice progression or recanalization of PVT.The patients are followed up every 2 months up to 18 month .Then statistical analysis will be done to find whether the Dabigatran is efficacious in cirrhotic patients for recanalization of PVT.

DETAILED DESCRIPTION:
Study population -All the patients of cirrhosis of liver patients visiting to ILBS and diagnosed to have non tumor portal vein thrombosis will be enrolled in the study.

Study Design - A Placebo Controlled Double Blinded RCT In this randomized controlled trial, the patients who satisfy the below inclusion and exclusion criteria will be included and they will be randomized, according to 2 groups (in total 84patients) to receive either Placebo or dabigatran 150 mg BD for 12months. These patients will be admitted to the hospital from OPD or emergency.

Study period - 1.5 years from ethics approval Intervention The patients in Group A will receive T. Dabigatran 150 mg twice a day .The patients in Group B will receive placebo [multivitamins] Monitoring and assessment At baseline, a complete history with clinical and physical examination, a record of demographic profile, standard of care biochemical investigations would be done. All included patients will be evaluated with -

1. Etiology of cirrhosis
2. Upper GI endoscopy
3. Haemogram (including reticulocyte count)
4. Coagulogram- PT/INR,APTT,TEG
5. Prothrombotic profile- protein c/protein-s/AT-III/Factor V Leiden mutation/ MTHFR C677T/PROTHROMBIN G20210A/ JAK2 V617F MUTATION / Anticardiolipin Ab.
6. Liver function tests, Renal function tests
7. Alpha fetoprotein/PIVKA II
8. USG abdomen with Doppler study
9. CECT-TP or CEMRI-TP to R/O HCC or angiography when PVT diagnosis doubtful.
10. HVPG+LIVER BIOPSY[optional]
11. Fibro scan
12. Child-Pugh score, MELD Subsequently, patients will be assessed clinically at the baseline and post-treatment every2 months till 18 months

Statistical Analysis:

The data collected will be analyzed using SPSS ver 22 by standard statistical analysis, were numerical data will be analyzed to find mean, median scores and categorical data will be analyzed using Chi square test and continuous data will be analyzed by student T test and any association will be analyzed by the univariate and multivariate analysis, log regression analysis along with ROC curve will be used and p<0.05 will be considered significant and results will be appropriately tabulated

Adverse Effects Hemorrhage - Fatal Major - intracranial, retroperitoneal, intraocular, muscle hematoma Minor TREATMENT IN CASE OF ADVERSE EFFECTS - Withdrawal of drug

Stopping rule of study Allergic reactions to drug Severe hemorrhage DIC Progression of PVT after 6 months viral reactivation leading to ACLF, acute hepatitis (viral, drug related, autoimmune flare), sepsis with severe coagulopathy

ELIGIBILITY:
Inclusion Criteria:

1. Clinical / radiological /histologic diagnosis of cirrhosis [Childs A&B - CTP<9]
2. Partial / total portal vein thrombosis (chronic)
3. Age- 18-70 years
4. Valid consent

Exclusion Criteria:

1. Age > 70 years
2. Presence of active infection (<2 weeks)
3. Use of anticoagulant drugs in the past 10 days
4. Pregnancy
5. HIV positivity
6. Recent (<7 days) transfusion with blood products.
7. History of bleeding in last 42 days
8. HCC / Other malignancy
9. Chronic kidney disease [ CrCl< 30]
10. Drug allergies
11. PVT with cavernoma formation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete recanalization of thrombus in both groups. | 1 year

SECONDARY OUTCOMES:
Number of participants with partial recanalization of thrombus in both groups. | 1 Year
Number of participants with improvements in Child-Turcotte-Pugh (CTP) in both groups. | 6 months
Number of participants with improvements in Child-Turcotte-Pugh (CTP) in both groups. | 1 year
Improvements in Model for End Stage Liver Disease (MELD) Score in both groups | 6 months
  MELD score ranges from 6 to 40.
Improvements in Model for End Stage Liver Disease (MELD) Score in both groups | 1 Year
  MELD score ranges from 6 to 40.
Number of participants with prevention of secondary decompensation in both groups | 1 Year
Adverse Events in both groups | 1 year
To study the changes in coagulation parameters by ROTEM(Rotational Thrombo Elastometry) analysis which includes CFT(clot formation time). | 6 Months
To study the changes in coagulation parameters by ROTEM(Rotational Thrombo Elastometry) analysis which includes CFT(clot formation time). | 12 Months
Number of participants with reduction in clinical complications in patients with PVT in both groups | 3 Months
Number of participants with reduction in clinical complications in patients with PVT in both groups | 6 Months
Number of participants with reduction in clinical complications in patients with PVT in both groups | 12 Months
To study the number of participants developing reoccurrence of PVT after treatment with Dabigatran for 12 months by Ultrasound Doppler of splenoportal venous system. | 12 months
To determine predictors for recurrence of PVT in patients with cirrhosis. | 1 year
To study the predictors of development of PVT in the population of cirrhosis patients screened who did not have PVT at the initiation of the study, for the development of new PVT over the period of the study | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided